CLINICAL TRIAL: NCT03152604
Title: The Effectiveness of a Pain Management Programme for Patients With Persistent Pain
Brief Title: Effectiveness of a Pain Management Programme
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Teesside University (Other)
Collaborators: South Tees Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, James Watson, PhD Student, Teesside University
Other Study IDs: 177/16
Record Dates: First submitted 2017-05-03; First posted 2017-05-15 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Persistent pain (PP) affects many people worldwide. Patient Education is central to good management. Pain neurophysiology education (PNE) is a new form of education. It aims to help patients 'reconceptualise' their understanding of pain away from the perception that PP is an indicator of tissue damage, to PP is due to a sensitised nervous system. This perception is considered a less threatening and more conducive to rehabilitation. There is a growing body of evidence supporting its effectiveness. One unpublished Australian study combined PNE with a pain management program and found significant beneficial effects. However, there is a need to test this intervention rigorously under randomised controlled trial conditions to inform clinical practice. The Medical Research Council state that during the development and evaluation of a complex intervention (in this case a PNE informed PMP), it is important to undertake feasibility work, to investigate the components of randomised controlled trial (RCT) methodology prior to a full scale trial. The overarching aim of this mixed-methods study is to develop a feasible research protocol for a RCT investigating the efficacy of a pain neurophysiology education informed pain management programme. In this feasibility study, participants with PP will be assessed before and after a PNE informed pain management program that they are due to receive as part of their usual care. In the week before the programme participants will attend Teesside University (TU) where they will complete a battery of outcome measures. A subsample of participants will also undergo a semi-structured interview. In the week following completion of their usual care PMP participants will once again attend TU where they will complete the same outcome measures and the same subsample of participants will undergo a second semi-structured interview. At this point participants will have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Have capacity to give informed consent
* 18+ years of age
* Have had pain that has persisted for greater than six months
* Have been referred to the pain management programme at James Cook University Hospital.

Exclusion Criteria:

* Pain arising from a non-musculoskeletal origin such as cancer pain, visceral pain or post stroke pain
* Have worsening neural signs
* Anyone being treated by or who has been treated by the researcher (JW)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with persistent musculoskeletal pain of greater than six months duration who have been referred to the pain management programme at James Cook University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2019-03-08 (Estimated); Study Completion 2019-03-08 (Estimated)

PRIMARY OUTCOMES:
The Brief Pain Inventory (Short Form) | Change from pre intervention (week 0) to post intervention (week 9)

SECONDARY OUTCOMES:
Centre of pressure | Change from pre intervention (week 0) to post intervention (week 9)
  Participants will be asked to stand quietly with your gaze at a fixation point, 3m away, at head height. When the participant has settled in double limb stance, arms by their sides they will be asked to instruct the researcher when they are ready. The centre of pressure data will then be recorded for 30 seconds. After the recording the participant will step off the force plate whilst it is re-calibrated giving them approximately one-minute rest before repeating the process so that three trials are recorded in total.
  The balance tests will then be repeated in the same way except participants will be instructed to close their eyes.
Fifty-foot walk at fastest speed | Change from pre intervention (week 0) to post intervention (week 9)
  Participants will be required to walk 25 feet, turn around and walk to the starting line as quickly as possible. The time taken will be recorded.
Repeated sit-to-stand | Change from pre intervention (week 0) to post intervention (week 9)
  Participants will be required to sit-to-stand from a standard chair 5 times as quickly as possible. The time taken will be recorded. This will be repeated a further time and the average time take for the two trials used for analysis to enhance reliability (Simmonds et al., 1998).
The Pain Catastrophising Scale | Change from pre intervention (week 0) to post intervention (week 9)
Neurophysiology of Pain Questionnaire | Change from pre intervention (week 0) to post intervention (week 9)
EQ-5D-5L | Change from pre intervention (week 0) to post intervention (week 9)
EQ-VAS | Change from pre intervention (week 0) to post intervention (week 9)
The Tampa Scale of Kinesiophobia | Change from pre intervention (week 0) to post intervention (week 9)
Pain Self-Efficacy Questionnaire | Change from pre intervention (week 0) to post intervention (week 9)
CORE-10 | Collected at the start of every session of the 8 session pain management programme which runs over 9 weeks
Stride Length | Change from pre intervention (week 0) to post intervention (week 9)
  It is measured on the line of progression between the heel points of two consecutive footprints of the same foot (left to left, right to right).
Step Length | Change from pre intervention (week 0) to post intervention (week 9)
  It is measured along the length of the walkway, from the heel center of the current footprint to the heel center of the previous footprint on the opposite foot.
H-H Base of Support or Base Width | Change from pre intervention (week 0) to post intervention (week 9)
  It is the vertical distance from heel center of one footprint to the line of progression formed by two footprints of the opposite foot.
Toe In / Toe Out | Change from pre intervention (week 0) to post intervention (week 9)
  It is the angle between the line of progression and the midline of the footprint. In Figure 7, theta is the angle between the mid-line of the right footprint and the line of progression. Angle theta is zero if the geometric mid- line of the footprint is parallel to the line of progression; positive, toe-out, when the mid-line of the footprint is outside the line of progression and negative, toe-in, when inside the line of progression. The unit of measure is degrees.
Step Width | Change from pre intervention (week 0) to post intervention (week 9)
  It is measured from the midline midpoint of the current footprint to the midline midpoint of the previous footprint on the opposite foot.
Stride width | Change from pre intervention (week 0) to post intervention (week 9)
  It is the vertical distance from midline midpoint of one footprint to the line formed by midline midpoints of two footprints of the opposite foot.
Step Time | Change from pre intervention (week 0) to post intervention (week 9)
  It is the time elapsed from first contact of one foot to first contact of the opposite foot. It is measured in seconds (sec).
Stride Time | Change from pre intervention (week 0) to post intervention (week 9)
  It is the time elapsed between the first contacts of two consecutive footfalls of the same foot. It is measured in seconds (sec).
Single Support | Change from pre intervention (week 0) to post intervention (week 9)
  It is the time elapsed between the Last Contact of the current footfall to the First Contact of the next footfall of the same foot.
% Single Support | Change from pre intervention (week 0) to post intervention (week 9)
  It is the % time elapsed between the Last Contact of the current footfall to the First Contact of the next footfall of the same foot.
Total Double Support | Change from pre intervention (week 0) to post intervention (week 9)
  The two periods when both feet are on the floor, are called initial double support and terminal double support. Initial double support occurs from heel contact of one footfall to toe-off of the opposite footfall. Terminal double support occurs from opposite footfall heel strike to support footfall toe-off. Total double support is the sum of the initial double support added to the terminal double support. It is measured in seconds (sec).
%Total Double Support | Change from pre intervention (week 0) to post intervention (week 9)
  The two periods when both feet are on the floor, are called initial double support and terminal double support. Initial double support occurs from heel contact of one footfall to toe-off of the opposite footfall. Terminal double support occurs from opposite footfall heel strike to support footfall toe-off. Total double support is the sum of the initial double support added to the terminal double support. It is measured in seconds (sec) and expressed as a percent of the Gait Cycle time for the same foot.
Stance Time | Change from pre intervention (week 0) to post intervention (week 9)
  The stance phase is the weight bearing portion of each gait cycle. It is initiated by heel contact and ends with toe off of the same foot. It is the time elapsed between the First Contact and the Last Contact of two consecutive footfalls on the same foot. It is also presented as a percentage of the Gait Cycle time.
% Stance Time | Change from pre intervention (week 0) to post intervention (week 9)
  The stance phase is the weight bearing portion of each gait cycle. It is initiated by heel contact and ends with toe off of the same foot. It is the time elapsed between the First Contact and the Last Contact of two consecutive footfalls on the same foot. It is presented as a percentage of the Gait Cycle time.
Swing Time | Change from pre intervention (week 0) to post intervention (week 9)
  It is initiated with toe off and ends with heel strike. It is the time elapsed between the Last Contact of the current footfall to the First Contact of the next footfall on the same foot. It is expressed in seconds (sec). The Swing Time is equal to the Single Support time of the opposite foot.
%Swing Time | Change from pre intervention (week 0) to post intervention (week 9)
  It is initiated with toe off and ends with heel strike. It is the time elapsed between the Last Contact of the current footfall to the First Contact of the next footfall on the same foot. It is expressed in seconds (sec) and it is presented as a percent of the Gait Cycle of the same foot. The Swing Time is equal to the Single Support time of the opposite foot.
Comfortable walking velocity | Change from pre intervention (week 0) to post intervention (week 9)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Teesside University, Middlesbrough, North Yorkshire
  - The Pain Clinic, South Tees Hospitals NHS Foundation Trust, Middlesbrough, North Yorkshire